CLINICAL TRIAL: NCT03538158
Title: A Personalized Health Behavior System to Promote Well-Being in Older Adults (FITTLE)
Brief Title: A Personalized Health Behavior System
Acronym: FITTLESenior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Florida Institute for Human and Machine Cognition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1806019352; R01AG053163 (NIH)
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Results first posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Social Isolation; Aging; Physical Activity
Keywords: Older adults; Physical well-being; Quality of life
MeSH Terms: conditions — Social Isolation; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention condition - Fittle Senior (Experimental): Participants will have access to the Fittle Senior System which will provide guided exercises and social support.
  Interventions: Behavioral: Intervention Condition
- Control condition - paper and pencil (Placebo Comparator): Participants will have a written booklet with exercises that they may do it on their own.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Intervention Condition — Participants will have access to Fittle Senior which will provide guided exercises and social support from other participants of the study.
  Arms: Intervention condition - Fittle Senior
Behavioral: Control Condition — Participants will have a paper booklet with suggested exercises that they may choose to complete for the duration of the study.
  Arms: Control condition - paper and pencil

SUMMARY:
The objectives of this study are to examine the usability and efficacy, for diverse older adults, of a new tablet-based dynamic system: the Fittle Senior System (FSS) that will provide: (1) personalized behavior-change programs for improved diet and increased physical activity and (2) online social interaction and support from small teams pursuing similar goals.

The proposed study involves a two group randomized trial where participants will be randomized to the Fittle Senior System or to a paper-based psycho-educational control condition following a baseline assessment. The duration of the intervention phase will involve an active 12-week intervention phase followed by a 12-week maintenance phase. We will recruit and randomize 180 community dwelling adults aged 65+ years, who live alone and are at risk for social isolation. Participants will be assessed at baseline, 3 months post active intervention and 3 months post maintenance (6 months following active intervention) on measures of health and health behaviors, and indices of social support.

DETAILED DESCRIPTION:
The proposed study will evaluate a new tablet-based dynamic system: the Fittle Senior System (FSS) that will provide: (1) personalized, goal-directed behavior-change programs for improved diet and increased physical activity and (2) online social interaction and support from small teams pursuing similar goals. The system builds on two technology-based systems developed by the investigative team: (1) the computer-based PRISM system (Czaja et al., 2015), designed for older populations to support social connectivity and well-being, and (2) the Fittle mobile platform (PARC) designed to support positive health behavior change through integrated online social support and personalized coaching based on artificial intelligence (AI). The Fittle program is based on Self-efficacy and Social Cognitive Theory (Bandura, 1998, 2001), Goal Setting (Locke & Latham, 2002) and the Theory of Planned Behavior (Ajzen, 1991). Fittle provides support for individuals and teams to progress through lifestyle challenges (e.g., poor eating habits, sedentary behavior), helping individuals master one health improving habit after another in a way that builds on previous achievements. Individuals choose from a variety of challenges to accomplish goals via an intelligent coaching agent and personalized, engaging user experiences. The objective is to maintain and reinforce perceived self-efficacy with daily goals that are perceived as being achievable, and to improve motivation and ability with goals that are perceived as not too easy. The program provides encouragement and social support through a team component. Thus, Fittle is designed to reinforce and build self-efficacy and positive attitudes.

ELIGIBILITY:
Inclusion Criteria:

* At least 60 years old
* Speak English
* Able to read at the 6th grade
* Plans to remain in the area for the study duration
* Pass TICS (Telephone Screen for Cognitive Status)

Exclusion Criteria:

* Cognitively impaired
* Visual or hearing impairment
* Actively engaged in structured physical exercise regularly
* Health conditions/illness that would affect participation

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara J. Czaja, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - University of Miami Miller School of Medicine, Miami, Florida
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with investigators upon request. This data will include sociodemographic data and outcome measures including SF-36, Loneliness Scale, Friendship Scale and Interpersonal Support Evaluation List (ISEL) scores. IPD will be free from any Personal Health Identifiers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available following the publication of the primary outcomes paper and will be available at request for 5 years.
Access Criteria: Data will be available to investigators at request.

REFERENCES:
- [Derived] Lieber SB, Moxley J, Mandl LA, Reid MC, Czaja SJ. Social support and physical activity: does general health matter? Eur Rev Aging Phys Act. 2024 Jun 20;21(1):16. doi: 10.1186/s11556-024-00347-6. PMID 38902616

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Condition - Fittle Senior | Control Condition - Paper and Pencil
Started | 92 | 89
12 Week Intervention Phase | 82 | 82
12 Week Maintenance Phase | 77 | 81
Completed | 77 | 81
Not Completed | 15 | 8
Not completed — Lost to Follow-up | 13 | 7
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Condition - Fittle Senior | Control Condition - Paper and Pencil | Total
Number analyzed (Participants) | 92 | 89 | 181
Age, Categorical [Count of Participants; unit: Participants] — Population: The number analyzed is different than the overall number of baseline participants because some participants were loss to follow up, withdrew from the study, or the data was not collected due to COVID-19.
  Participants
    number analyzed (Participants) | 87 | 88 | 175
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 17 | 17 | 34
    >=65 years | 70 | 71 | 141
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number analyzed is different than the overall number of baseline participants because some participants were loss to follow up, withdrew from the study, or the data was not collected due to COVID-19.
  Participants
    number analyzed (Participants) | 89 | 87 | 176
    Female | 74 | 67 | 141
    Male | 15 | 20 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number analyzed is different than the overall number of baseline participants because some participants were loss to follow up, withdrew from the study, or the data was not collected due to COVID-19.
  Participants
    number analyzed (Participants) | 89 | 88 | 177
    Hispanic or Latino | 12 | 12 | 24
    Not Hispanic or Latino | 77 | 76 | 153
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 72 | 74 | 146
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 4 | 1 | 5
VO2 Max [Mean (Standard Deviation); unit: mL/kg/min] — Population: The number analyzed is different than the overall number of baseline participants because some participants were loss to follow up, withdrew from the study, or the data was not collected due to COVID-19.
  mL/kg/min
    number analyzed (Participants) | 46 | 41 | 87
    (all) | 16.6 (5.4) | 16.8 (4.9) | 16.7 (5.4)
Timed Up and Go [Mean (Standard Deviation); unit: Seconds] — To start the TUG, you will sit in the chair with your arms resting comfortably on your lap or at your sides.
  The test begins when the therapist says "Go" and starts the stopwatch. You would then be timed as you rise from the chair, walk three meters, turn around, return to the chair, and sit down.
  The recorded time on the stopwatch is the TUG score.
  Measure to assess mobility. A faster time indicates a better functional performance.
  An older adult who takes ≥12 seconds to complete the TUG is at risk for falling. Population: The number analyzed is different than the overall number of baseline participants because some participants were loss to follow up, withdrew from the study, or the data was not collected due to COVID-19.
  Seconds
    number analyzed (Participants) | 56 | 50 | 106
    (all) | 10.5 (3) | 10.2 (2.6) | 10.4 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: VO2 Max
Description: Higher score of VO2 max indicates more oxygen consumption during incremental exercise.
Time Frame: Baseline, 3 month follow-up and 6 month follow-up
Population: The number analyzed is different than the number of subjects in the participant flow because some participants were loss to follow up, withdrew from the study, or the data was not collected due to COVID-19.
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Intervention Condition - Fittle Senior | Control Condition - Paper and Pencil
Number analyzed (Participants) | 46 | 41
mL/kg/min
  Baseline | 16.6 (5.4) | 16.8 (4.9)
  3 month follow-up: number analyzed (Participants) | 27 | 16
  3 month follow-up | 15.7 (4.4) | 18.5 (5.6)
  6 month follow-up: number analyzed (Participants) | 2 | 4
  6 month follow-up | 20.2 (1.4) | 17.3 (2)
Statistical Analysis 1: Comparison: Intervention Condition - Fittle Senior vs Control Condition - Paper and Pencil; Test type: Superiority; p = .82, Mixed Models Analysis; F(2,131)=.07; Slope = 5.7, 95% CI 2-sided [-287.7 to 299.1]

2. Secondary Outcome: Timed Up and Go
Description: To start the TUG, you will sit in the chair with your arms resting comfortably on your lap or at your sides.
  The test begins when the therapist says "Go" and starts the stopwatch. You would then be timed as you rise from the chair, walk three meters, turn around, return to the chair, and sit down.
  The recorded time on the stopwatch is the TUG score. Measure to assess mobility. A faster time indicates a better functional performance.
  An older adult who takes ≥12 seconds to complete the TUG is at risk for falling.
Time Frame: Baseline, 3 month follow-up and 6 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Intervention Condition - Fittle Senior | Control Condition - Paper and Pencil
Number analyzed (Participants) | 56 | 50
Seconds
  Baseline | 10.5 (3) | 10 (2.6)
  3 Month Follow-Up: number analyzed (Participants) | 26 | 12
  3 Month Follow-Up | 9.2 (1.8) | 8.6 (3.9)
  6 Month Follow-Up: number analyzed (Participants) | 3 | 4
  6 Month Follow-Up | 10 (2.3) | 8.6 (1.1)
Statistical Analysis 1: Comparison: Intervention Condition - Fittle Senior vs Control Condition - Paper and Pencil; Test type: Superiority; p = .97, Mixed Models Analysis; F(2,75)=.03; Slope = .5, 95% CI 2-sided [-3.5 to 4.4]

3. Other Pre Specified Outcome: Change in Functional Health and Well-being as Measured by Modified SF-36
Description: Higher score means better functional health and well-being. Range (0-1400)
Time Frame: Baseline, 3 month follow-up and 6 month follow-up
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Loneliness as Measured by Loneliness Scale
Description: Higher score indicates a greater degree of loneliness. Range (0-80)
Time Frame: Baseline, 3 month follow-up and 6 month follow-up
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Social Isolation as Measured by Friendship Scale
Description: Measures the level of social isolation. Lower score indicates less social isolation. Range (0-24)
Time Frame: Baseline, 3 month follow-up and 6 month follow-up
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Social Support as Measured by Interpersonal Support Evaluation List - ISEL
Description: Measures the level of functional social support. Higher scores indicates better and more social support
Time Frame: Baseline, 3 month follow-up and 6 month follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The 6 months the participant was enrolled in the study.
Arm/Group | Intervention Condition - Fittle Senior | Control Condition - Paper and Pencil
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/89
Serious Adverse Events (participants affected / at risk) | 3/92 | 3/89
Other Adverse Events (participants affected / at risk) | 4/92 | 5/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Condition - Fittle Senior (N=92) | Control Condition - Paper and Pencil (N=89)
Heart surgery (Cardiac disorders) | 0 (0) | 1 (1)
Cancer (General disorders) | 2 (2) | 0 (0)
Kidney Stone (Renal and urinary disorders) | 1 (1) | 0 (0)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Kidney Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Condition - Fittle Senior (N=92) | Control Condition - Paper and Pencil (N=89)
Fall (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Shoulder Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/58/NCT03538158/Prot_SAP_000.pdf